CLINICAL TRIAL: NCT05084443
Title: Effect of Roselle-based Drink on Blood Pressure, Antioxidative Activity and Skin Condition
Brief Title: Effect of Roselle-based Drink on Blood Pressure and Skin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chung Shan Medical University (Other)
Responsible Party: Principal Investigator, Chin Kun Wang, Professor, Chung Shan Medical University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: CS11102
Record Dates: First submitted 2021-09-29; First posted 2021-10-19 (Actual); Last update posted 2021-10-26 (Actual); Status verified 2021-10

CONDITIONS: Other Skin and Subcutaneous Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo/Control (Placebo Comparator): Placebo drink-- Orally (200 ml/day)
  Interventions: Dietary Supplement: Drink
- Roselle Based drink (Test) (Experimental): Roselle-Based Drink--- Orally (200 ml/day)
  Interventions: Dietary Supplement: Drink

INTERVENTIONS:
Dietary Supplement: Drink — Roselle and placebo drink for 6 months
  Other Names: Roselle Drink (SF-R product of Han Bu)

SUMMARY:
This randomized, placebo-controlled, double-blind, and cross-over study was designed to check whether the roselle-based drink (2 bottles every day) can alter blood pressure and skin condition in elderly healthy subjects.

DETAILED DESCRIPTION:
The subjects were assigned into two groups (control group and test group), each group subject was requested to drink 2 bottles every day (100 mL/bottle, one in the morning and another in the evening), the rate of drinking is 75.42%. There are 39 subjects (25 females and 14 males) completely involved in the thirteen-month trial (cross-over). Blood samples were collected at the initial, 3rd, 6th, 7th, 10th, 13th months of the trial. Skin examinations were performed at the initial, 6th, 7th, 13th months.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults
* Subjects should not be under any medication
* Subject must be able to drink

Exclusion Criteria:

* Subjects with chronic renal, liver or cardiac disorders, Diabetes, hyperlipidemia.
* Also pregnant women, chain smokers, high alcohol consumers should not be included.

Ages: 40 Years to 81 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2017-09-11 (Actual); Primary Completion 2018-06-15 (Actual); Study Completion 2018-10-19 (Actual)

PRIMARY OUTCOMES:
Blood pressure by sphygmomanometer (mmHg) | 6 months
  Both systolic and diastolic blood pressure were changed after Roselle drink

CONTACTS AND LOCATIONS:
Overall Officials: Chin-Kun Wang, Ph.D, Principal Investigator — Chung Shan Medical University
Locations (1):
- Chung Shan Medical University, Taichung, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No